CLINICAL TRIAL: NCT02416570
Title: Is Clarithromycin a Potential Treatment for Cachexia in People With Lung Cancer?
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At 6 months 1 participant recruited. Study deemed not feasible and discontinued.
Sponsor: University of Nottingham (Other)
Collaborators: Roy Castle Lung Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 14102
Record Dates: First submitted 2015-03-06; First posted 2015-04-15 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Cachexia; Lung Cancer
Keywords: Clarithromycin
MeSH Terms: conditions — Cachexia; Lung Neoplasms | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarithromycin (Active Comparator): Clarithromycin 250mg by mouth twice a day for 8 weeks
  Interventions: Drug: Clarithromycin
- Placebo (Placebo Comparator): Placebo matched capsule one capsule by mouth twice a day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clarithromycin
  Arms: Clarithromycin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study aims to identify if clarithromycin (CLM) has potential as a widely available and inexpensive treatment for cachexia (the loss of muscle mass) in people with non-small cell lung cancer (NSCLC). Half the participants will receive clarithromycin and half will receive a placebo.

DETAILED DESCRIPTION:
Clarithromycin has been reported to significantly improve markers of inflammation, body weight, need for hospital admission and survival in 42 patients with NSCLC. Compared to patients receiving best supportive care only, those receiving Clarithromycin had an improved median survival of ~8 months (535 vs. 277 days), stayed at home longer (439 vs. 139 days) and reported no adverse effects.

In another study, 33 patients with NSCLC were given Clarithromycin for 3 months and compared to a matched control group there was a reduction in IL-6 levels which correlated with an improvement in body weight (gain 4 vs. 1kg) and survival. Thus, by reducing inflammation, Clarithromycin may be impeding the cachectic process, preserving body weight, physical function and independence and increasing survival.

These studies of Clarithromycin in NSCLC have limitations, e.g. lack of placebo-control, no direct assessment of lean body mass.

This feasibility study will obtain data to inform the viability and design of a larger randomised, double-blind, placebo-controlled, phase III study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stage IV, pathologically confirmed, NSCLC not suitable for/declining/not tolerating 1st/2nd-line palliative chemotherapy, or following completion of 1st/2nd-line palliative chemotherapy
* A likely prognosis of ≥3 months.
* Cachexia on the basis of any of the following, weight loss >5% over past 6 months, or BMI <20kg/m2 and weight loss >2%, or appendicular skeletal muscle index determined by duel energy x-ray absorptiometry consistent with sarcopenia and weight loss >2%.
* Systemic inflammation on the basis of a C-reactive protein >10mg/L.
* Adequate renal function as defined by creatinine ≤132micromol/L and eGFR ≥30mL/min/1.73m2
* Adequate liver function as defined by the following parameters, bilirubin ≤25micromol/L, and AST and ALT ≤2 times upper limit of normal, unless liver metastases, in which case ≤5 times upper limit of normal
* Prepared to suspend, if necessary, the use of certain statins and/or substitute the use of domperidone for an alternative anti-emetic for the duration of the study

Exclusion Criteria:

* ECOG Performance Status 3 or 4
* Little or no food intake
* Weight loss >10% in 1 month or >20% in total
* Known hypersensitivity to clarithromycin
* Inability to accurately measure QT interval, e.g. atrial fibrillation
* QTc prolongation >450 milliseconds in a male, or 470 milliseconds in a female
* History of ventricular arrhythmia
* Severe cardiac insufficiency (NYHA class >2)
* Untreated hypokalaemia/hypomagnesaemia
* Active infection requiring antibiotics
* Current or recent (within last 4 weeks) history of Clostridium difficile, eating disorder, dysphagia, malabsorption or diarrhoea
* Untreated adrenal or thyroid diseases
* Brain metastases
* Use of corticosteroids/progestogens
* Use of chemotherapy, other immunosuppressive, or antiviral (e.g. hepatitis C, HIV) drugs within 4 weeks
* Drugs which are contra-indicated (except certain statins which can be temporarily suspended and domperidone which can be substituted for an alternative anti-emetic) or should be avoided in patients receiving clarithromycin, either because of the risk of a drug-drug interaction and/or prolonged QT
* Pregnancy
* Breast Feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of a phase 3 study | 1 year
  The number of patients recruited to the study as a measure of feasibility.

SECONDARY OUTCOMES:
Tolerability of clarithromycin | 1 year
  Number of patients taking >80% of prescribed doses as a measure of tolerability.
Safety of clarithromycin | 1 year
  Number of adverse events as a measure of safety.
Safety of clarithromycin | 1 year
  Number of patients with prolongation of the QT interval as a measure of safety.
Effect of clarithromycin | 1 year
  Change from baseline in body composition at 8 weeks as a measure of effect.
Effect of clarithromycin | 1 year
  Change from baseline in hand grip strength at 8 weeks as a measure of effect.
Effect of clarithromycin | 1 year
  Change from baseline in 5 repetition sit to stand test speed at 8 weeks as a measure of effect.
Effect of clarithromycin | 1 year
  Change from baseline in 4 metre gait speed at 8 weeks as a measure of effect.
Effect of clarithromycin | 1 year
  Change from baseline in EQ-5D-5L at 8 weeks as a measure of effect.
Effect of clarithromycin | 1 year
  Change from baseline in QLC Q30 at 8 weeks as a measure of effect.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilcock, Principal Investigator — University of Nottingham